CLINICAL TRIAL: NCT05469282
Title: A Single Center Clinical Trial to Evaluate the Efficacy and Safety of Blood Circulation Improvement Using an Investigational Medical Device (Model Name CGM MB-1701) for the Risk Group of Deep Vein Thrombosis (DVT) and the Ordinary Person
Brief Title: CEFID-I (CEra Flow Improves DVT-1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceragem Clinical Inc. (Industry)
Responsible Party: Sponsor
Organization: Ceragem Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-06-043
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Blood Circulation Disorder; Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood circulation treatment (Experimental): Blood circulation treatment for the risk group for Deep Vein Thrombosis (DVT) and the ordinary person
  Interventions: Device: Blood circulation device

INTERVENTIONS:
Device: Blood circulation device — Blood circulation device of CGM MB-1701 (Ceragem Master V6)

SUMMARY:
The study is a single center clinical trial to evaluate the efficacy and safety of blood circulation improvement using an investigational medical device, which is a product on the market and it's name is Ceragem Master V6, for the risk group of Deep Vein Thrombosis (DVT) and the ordinary person. The study compares before and after the application by one time application.

DETAILED DESCRIPTION:
The efficacy and safety evaluation are conducted before and after (or during) the application of the test device. The investigator shall apply an investigational device once when visiting a suitable subject for one day.

ELIGIBILITY:
Inclusion Criteria for all subjects; 1. Adult men and women over 19 years of age 2. Subjects who have not been diagnosed with deep vein thrombosis in the lower extremities through the following test results prior to the application of medical devices.

1. Subjects diagnosed by Doppler ultrasonography as having no blood clots in the femoral vein and the vena poplitea
2. D-dimer negative test result (Even if the D-dimer test is positive, the subject can be selected through the additional test at the discretion of investigator.)

3. Subjects who fully understand the purpose and procedure of the study and wish to participate in clinical trials with voluntary consent

Additional Inclusion Critetia for the DVT risk subjects;

1. Subjects have two or more points of venous thromboembolism (hereinafter referred to as VTE) clinical prediction score (Two-level wells scroe) at the time of screening

Exclusion Criteria:

1. Subjects who complain of a decrease in the sensation of the lower extremities or who is unable to feel the sensation of pain
2. Subjects who have inflammation or trauma on the skin that directly touches the device

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity (PSV) change | While 2 consecutive application (36 minutes) per one subject
  Evaluate the maximum blood flow rate (PSV) change in the femoral vein when applied compared to before application of the device using ultrasonic at Visit 1

SECONDARY OUTCOMES:
Antero-posterior (AP) diameter | While 2 consecutive application (36 minutes) per one subject
  Evaluate the the maximum AP diameter change of the femoral vein when applied compared to before the device is applied using ultrasonic at Visit 1.
Cross Sectional Area | While 2 consecutive application (36 minutes) per one subject
  Evaluate the maximum CSA area change of the femoral vein when applied compare to before the device is applied using ultrasonic at Visti 1.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Soon Yoon, MD, Principal Investigator — Presbyterian medical center
Locations (1):
- Presbyterian Medical Center, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided